CLINICAL TRIAL: NCT02373735
Title: Effect of Stroke Volume Variation Guided Fluid Therapy on the Blood Loss and Postoperative Outcomes in Radical Cystectomy
Brief Title: Effect of SVV Guided Fluid Therapy on Blood Loss and Postoperative Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S2014-2192
Record Dates: First submitted 2015-02-12; First posted 2015-02-27 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Bladder Cancer
Keywords: stroke volume variation; radical cystectomy; blood loss; postoperative complications
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hemorrhage; Postoperative Complications | interventions — Crystalloid Solutions; Ringer's Lactate; Colloids; Mannitol; Furosemide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (SVV <10% group) (Active Comparator): * infuse crystalloid (Hartmann's solution) 6-10 ml/kg/hr continuously during surgery
  * infuse colloid (Volulyte) 200 ml if SVV is ≥ 10% during the surgery
  Interventions: crystalloid (Hartmann's solution), colloid (Volulyte)
  Interventions: Other: crystalloid; Other: colloid
- Group B (SVV 10-20% group) (Experimental): * infuse crystalloid (Hartmann's solution) 2-4 ml/kg/hr until cystectomy, 6-10 ml/kg/hr after cystectomy
  * infuse colloid (Volulyte) 200 ml if SVV is > 20%
  * infuse mannitol 0.5 g/kg or lasix 5 mg if SVV < 10%
  Interventions: crystalloid (Hartmann's solution), colloid (Volulyte), mannitol, lasix
  Interventions: Other: crystalloid; Other: colloid; Other: mannitol; Other: lasix

INTERVENTIONS:
Other: crystalloid — Group A (SVV <10%): infuse crystalloid 6-10 ml/kg/hr during surgery. Group B (SVV 10-20%): infuse crystalloid 2-4 ml/kg/hr until cystectomy, 6-10 ml/kg/hr after cystectomy
  Other Names: Hartmann's solution
Other: colloid — Group A (SVV <10%): infuse colloid 200 ml if SVV is ≥ 10%. Group B (SVV 10-20%): infuse colloid 200 ml if SVV is > 20%
  Other Names: volulyte
Other: mannitol — Group B (SVV 10-20%): infuse mannitol 0.5 g/kg if SVV is < 10%
  Arms: Group B (SVV 10-20% group)
Other: lasix — Group B (SVV 10-20%): infuse lasix 5 mg if SVV is < 10%
  Arms: Group B (SVV 10-20% group)

SUMMARY:
The purpose of this study is to investigate the effect of stroke volume variation (SVV) guided fluid therapy on the blood loss and postoperative outcomes in radical cystectomy.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of stroke volume variation(SVV) guided fluid therapy on the blood loss and postoperative outcomes in radical cystectomy. Patients were randomized to fluid management to maintain <10% SVV (group A), or to undergo fluid management during radical cystectomy to maintain SVV 10-20% (group B). Intraoperative blood loss and hemodynamic parameters, perioperative laboratory data, and postoperative complications were compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer patients who received radical cystectomy
* Patients with American Society of Anesthesiologists physical status scale classification 1, 2
* Patients who agree with written informed consent

Exclusion Criteria:

* Patients with history of arrhythmia, heart failure patients
* Patients with history of renal failure patients
* Patients with history of abdominal surgery
* Patients who received emergency operation
* Patients who do not agree with study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | During operation

SECONDARY OUTCOMES:
Postoperative complications (cardiovascular complications, gastrointestinal complications, pulmonary complications, renal complications, infection, death) | During 30 days after operation
  Postoperative complications include cardiovascular complications, gastrointestinal complications, pulmonary complications, renal complications, infection, death
Length of hospital stay/ICU stay | participants will be followed for the duration of hospital stay, an expected average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, M.D., Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea